CLINICAL TRIAL: NCT01797289
Title: The Prevalence of Pulmonarym Embolism in Patients With the First Episode of Syncope
Brief Title: Prevalence of Pulmonary Embolism in Patients With Syncope
Acronym: PESY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Paolo Prandoni, Professor, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 52823P
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Syncope; Pulmonary Embolism
Keywords: syncope; pulmonary embolism
MeSH Terms: conditions — Syncope; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- First episode of loss of consciousness (Experimental)
  Interventions: Other: Lung CT or V/Q scanning in patients with a high pre-test clinical probability of PE and/or a positive D-dimer

INTERVENTIONS:
Other: Lung CT or V/Q scanning in patients with a high pre-test clinical probability of PE and/or a positive D-dimer

SUMMARY:
All patients consecutively referred with the first episode of transient and short-lasting loss of consciousness will have a diagnostic workup for the assessment of the most common causes of syncope, and will be evaluated for the presence of pulmonary embolism (PE) with the use of an internationally accepted algorithm including a pre-test clinical probability (PTP according to the method of Wells et al.) and a high-sensitivity quantitative D-dimer assay. If the PTP is low and D-dimer negative, PE will be excluded. All other patients will undergo confirmatory diagnostic tests (either computerized tomography or ventilation/perfusion lung scanning) in order to confirm or rule out the presence of PE.

ELIGIBILITY:
Inclusion Criteria:

* first episode of syncope

Exclusion Criteria:

* previous episodes of syncope
* ongoing anticoagulation
* age younger than 18 years
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2012-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To assess the prevalence of PE in a large series of consecutive patients presenting with the first episode of syncope | Up to 48 hours after hospital admission

SECONDARY OUTCOMES:
To assess the prevalence of pulmonary embolism in patients with apparently unexplained syncope | Up to one week after hospital admission

OTHER OUTCOMES:
To assess the prevalence of pulmonary embolism in patients with syncope with a high pre-test probability of PE and/or a positive D-dimer | Up to 48 hours after admission

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Medica 2 University of Padua, Padua, Italy

REFERENCES:
- [Derived] Prandoni P, Lensing AW, Prins MH, Ciammaichella M, Perlati M, Mumoli N, Bucherini E, Visona A, Bova C, Imberti D, Campostrini S, Barbar S; PESIT Investigators. Prevalence of Pulmonary Embolism among Patients Hospitalized for Syncope. N Engl J Med. 2016 Oct 20;375(16):1524-1531. doi: 10.1056/NEJMoa1602172. PMID 27797317